CLINICAL TRIAL: NCT01553565
Title: Prospective Comparison of Cold Polypectomy and Conventional Polypectomy for Small Colorectal Polyps in Patients Taking Antithrombotic Agents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Showa Inan General Hospital (Other)
Responsible Party: Principal Investigator, Akira Horiuchi, Chief, Digestive Disease Center, Showa Inan General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: cold vs.hot
Record Dates: First submitted 2012-03-10; First posted 2012-03-14 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Colorectal Polyps
Keywords: 10 mm in diameter; antithrombotic agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional polypectomy (Active Comparator): All colorectal polyps up to 10 mm found except for tiny hyperplastic polyps in the rectum and distal sigmoid colon are removed with electrocautery. Submucosal injection of some solution before the removal are not performed.
  Interventions: Procedure: Cold polypectomy
- Cold polypectomy (Experimental)
  Interventions: Procedure: Cold polypectomy

INTERVENTIONS:
Procedure: Cold polypectomy — All colorectal polyps up to 10 mm found except for tiny hyperplastic polyps in the rectum and distal sigmoid colon are removed. The technique is cold resection of the polyp without tenting and then suction of the transected polyp into a trap followed by submission to histopathological evaluation.
  Other Names: Cold snare polypectomy

SUMMARY:
1. Background: The ideal method to remove small colorectal polyps in patients who are taking antithrombotic agents is unknown.
2. Aim: The aim of this study is to evaluate postpolypectomy bleeding and the complete retrieval rate after the removal by colon snare transection without electrocautery for small polyps in patients who are taking antithrombotic agents.
3. Design: A prospective, consecutive study.
4. Setting: Municipal hospital outpatients.
5. Interventions: Polypectomy by cold snare technique (Cold polypectomy) was performed for colorectal polyps up to 10 mm in diameter in patients who continue to take antithrombotic agents. The primary outcome measure was bleeding within two weeks after polypectomy. Secondary outcome measure was the complete retrieval rate of colorectal polyps based on the pathological examination.

ELIGIBILITY:
Inclusion Criteria:

* Patients with colorectal polyps up to 10 mm in diameter. The patients continue to take antithrombotic agents.

Exclusion Criteria:

* patients are less than 20 years old,
* pregnant,
* American Society of Anesthesiologists class III and IV,
* overweight (body weight > 100 kg), or
* allergic to propofol used or its components (soybeans or eggs),
* with previous colorectal surgical resection.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Postpolypectomy bleeding | 2 weeks
  Bleeding within two weeks after polypectomy

SECONDARY OUTCOMES:
Complete retrieval rate of colorectal polyps | 2 weeks
  The complete retrieval rate of colorectal polyps based on the pathological examination.

CONTACTS AND LOCATIONS:
Overall Officials: Akira Horiuchi, MD, Principal Investigator — Showa Inan General Hospital
Locations (1):
- Showa Inan General Hospital, Komagane, Nagano, Japan

REFERENCES:
- [Derived] Horiuchi A, Nakayama Y, Kajiyama M, Tanaka N, Sano K, Graham DY. Removal of small colorectal polyps in anticoagulated patients: a prospective randomized comparison of cold snare and conventional polypectomy. Gastrointest Endosc. 2014 Mar;79(3):417-23. doi: 10.1016/j.gie.2013.08.040. Epub 2013 Oct 11. PMID 24125514